CLINICAL TRIAL: NCT02078388
Title: Correlation Between Genetic Variants and Long-term Cardiac Effects Induced by Doxorubicin in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Haematology-Oncology, Lee Soo Chin, National University Hospital, Singapore
Other Study IDs: 2013/01090
Record Dates: First submitted 2013-12-08; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer,Doxorubicin: Breast cancer patients who received at least one cycle of doxorubicin-containing adjuvant chemotherapy for treatment of early stage breast cancer at least 12 months ago and who had a pre-doxorubicin echocardiography done at NUHS will be enrolled. Study subjects will donate one sample of blood (20ml) for genetic and biomarker studies related to breast cancer and anthracyclines pharmacodynamics. An echocardiography will be performed to measure left ventricular ejection fraction, and compared with the subject's pre-doxorubicin echocardiography done at NUH. Correlative analysis will be performed between genetic variants and left ventricular ejection change.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin

SUMMARY:
The purpose of this study is to identify the genetic variants that are associated with higher risk of doxorubicin-induced cardiotoxicity can contribute towards developing a predictive algorithm comprising both clinical and genetic factors to select patients who should avoid treatment with anthracyclines.

Hypothesis of this study is certain functional variants in genes that encode for metabolizing enzymes and/or targets in the doxorubicin pharmacology pathway may increase the risk of doxorubicin-induced cardiomyopathy

DETAILED DESCRIPTION:
Doxorubicin is one of the cornerstone therapies in adjuvant chemotherapy in early stage breast cancer. Cumulative doses of 240mg/m2 (4 cycles of doxorubicin/cyclophosphamide) and 300mg/m2 (6 cycles of doxorubicin/cyclophosphamide) are typically administered in the adjuvant setting, which is associated with <1% chance of severe cardiotoxicity, and are thus considered 'safe dose ranges'. However, Blanco et al recently reported childhood cancer survivors with the CBR3 (a metabolizing enzyme of doxorubicin) V244M homozygous G genotypes to be at increased risk of cardiomyopathy following exposure to anthracyclines doses as low as 101-150mg/m2, suggesting that there is no safe dose threshold for individuals with certain genotypes. We have previously studied several genes in the doxorubicin pharmacology pathway, including CBR1, CBR3, and AKR1C3, and found correlation between functional variants in CBR3 and AKR1C3 with doxorubicin-induced myelosuppression. The CBR3 G allele is present in about 50-60% of the Singapore population, and we postulate that these common variants may similarly modify the risk of anthracyclines-induced cardiomyopathy in adult breast cancer patients. Post-treatment echocardiography is not routinely performed in patients who complete adjuvant anthracyclines-containing chemotherapy. We believe that some of these high-risk individuals may have subclinical reduced left ventricular ejection fraction that may in the future increase the risk of congestive cardiac failure in the presence of other risk factors (eg hypertension, anemia, serious infection, etc). Identifying these individuals could therefore be important as early treatment with ACE inhibitors may improve cardiac function. Confirming the correlation between genetic variants including the CBR3 V244M can also help to develop a predictive algorithm in the future to identify patients in whom anthracyclines should be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 21 years
* Signed informed consent from patient or legal representative.

Exclusion Criteria:

* Pregnancy
* Breast feeding.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who received at least one cycle of doxorubicin-containing adjuvant chemotherapy for treatment of early stage breast cancer at least 12 months ago and who had a pre-doxorubicin echocardiography done at NUHS will be enrolled.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change the functional variants in genes involved in doxorubicin pharmacology with doxorubicin-induced cardiomyopathy in adult breast cancer survivors. | 1 year
  Identification of genetic variants that are associated with higher risk of doxorubicin-induced cardiotoxicity can contribute towards developing a predictive algorithm comprising both clinical and genetic factors to select patients who should avoid treatment with anthracyclines.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Blanco JG, Sun CL, Landier W, Chen L, Esparza-Duran D, Leisenring W, Mays A, Friedman DL, Ginsberg JP, Hudson MM, Neglia JP, Oeffinger KC, Ritchey AK, Villaluna D, Relling MV, Bhatia S. Anthracycline-related cardiomyopathy after childhood cancer: role of polymorphisms in carbonyl reductase genes--a report from the Children's Oncology Group. J Clin Oncol. 2012 May 1;30(13):1415-21. doi: 10.1200/JCO.2011.34.8987. Epub 2011 Nov 28. PMID 22124095
- [Background] Fan L, Goh BC, Wong CI, Sukri N, Lim SE, Tan SH, Guo JY, Lim R, Yap HL, Khoo YM, Iau P, Lee HS, Lee SC. Genotype of human carbonyl reductase CBR3 correlates with doxorubicin disposition and toxicity. Pharmacogenet Genomics. 2008 Jul;18(7):621-31. doi: 10.1097/FPC.0b013e328301a869. PMID 18551042